CLINICAL TRIAL: NCT03158194
Title: Cognitive Behavior Therapy for Anxiety-related Asthma in Adults.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Catarina Almqvist Malmros, Professor, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MANTRA 01
Record Dates: First submitted 2017-05-16; First posted 2017-05-18 (Actual); Last update posted 2018-03-08 (Actual); Status verified 2018-03

CONDITIONS: Asthma
Keywords: Anxiety; Stress; Asthma
MeSH Terms: conditions — Asthma; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Single-subject multiple baseline design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CBT for anxiety-related asthma (Experimental): Ten to twelve weekly sessions of CBT targeting enhanced function and decreased symptoms of anxiety.
  Interventions: Behavioral: CBT for anxiety-related asthma

INTERVENTIONS:
Behavioral: CBT for anxiety-related asthma — The specific assignments in the intervention will be based on individual behavior analysis for each participant.

SUMMARY:
This is a study to develop a protocol on Cognitive behavior therapy (CBT) for asthma-related anxiety that in a consecutive study can be translated to internet-delivered CBT.

DETAILED DESCRIPTION:
Asthma is one of the most common chronic diseases around the world, with a high prevalence of anxiety disorders. Cognitive behaviour therapy (CBT) has been shown to increase psychological well-being for anxiety-related asthma. Our primary aim is to develop a standardized CBT protocol for asthma-related anxiety that can be transferred to internet-delivered CBT. Ten participants will be included in a single-subject multiple baseline design. They will all receive 10-12 sessions of CBT.

ELIGIBILITY:
Inclusion Criteria:

* asthma diagnosed by a physician
* anxiety or stress related to asthma

Exclusion Criteria:

* severe psychiatric disorder (e.g. psychotic disorder, addiction disorder, suicidal ideation).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-08-16 (Actual); Primary Completion 2018-03-07 (Actual); Study Completion 2018-03-07 (Actual)

PRIMARY OUTCOMES:
Penn State Worry Questionnaire | Baseline to 12 weeks
  Change in subjective worry measured with a self-rating scale weekly during 1-3 weeks at baseline and at 10 to 12 weeks post treatment for analysis of effect.

SECONDARY OUTCOMES:
Anxiety Sensitivity Index-3 | Baseline to 12 weeks
  Change in anxiety sensitivity measured with a self-rating scale weekly during 1-3 weeks at baseline and at 10 to 12 weeks post treatment for analysis of effect.
Short Health Anxiety Inventory (SHAI) | Baseline to 12 weeks
  Change in health anxiety measured with a self-rating scale weekly during 1-3 weeks at baseline and at 10 to 12 weeks post treatment for analysis of effect.
Asthma Quality of Life Questionnaire | Baseline to 12 weeks
  Change in asthma-related quality of life measured with a self-rating scale at pretreatment and at 10 to 12 weeks post treatment for analysis of effect.
Asthma control test | Baseline to 12 weeks
  Change in asthma control measured with a self-rating scale daily during weekly 1-3 weeks at baseline and at 10 to 12 weeks post treatment for analysis of effect.
Catastrophizing about asthma Scale | Baseline to 12 weeks
  Change in catastrophizing cognitions about asthma measured with a self-rating scale weekly during 1-3 weeks at baseline and at 10 to 12 weeks post treatment for analysis of effect.
Perceived Stress Scale | Baseline to 12 weeks
  Change in perceived stress measured with a self-rating scale weekly 1-3 weeks at baseline and at 10 to 12 weeks post treatment for analysis of effect.
Patient Health Questionnaire | Baseline to 12 weeks
  Change in depression measured with a self-rating scale at baseline and at 10 to 12 weeks post treatment for analysis of effect.

CONTACTS AND LOCATIONS:
Overall Officials: Catarina Almqvist Malmros, MD, PhD, Principal Investigator — Department of Medical Epidemiology and Biostatistics, Karolinska Institutet
Locations (1):
- Department of Medical Epidemiology and Biostatistics, Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No